CLINICAL TRIAL: NCT03676686
Title: A Prospective Single-arm Investigation to Assess the Efficacy, of Topical "Nåva" Foot Cream for 8 Weeks of Treatment in Patients With Mild to Moderate Tinea Pedis Interdigitalis and Heal Cracks, Calluses and/or Dry Feet.
Brief Title: Study With Nåva Foot Cream in Patients With Tinea Pedis Interdigitalis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natumin Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nåva Foot Cream_1
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nåva Foot Cream (Experimental): Topical Nåva foot cream administered twice daily.
  Interventions: Device: Nåva Foot Cream

INTERVENTIONS:
Device: Nåva Foot Cream — Nåva Foot Cream is a Medical device (EU class IIa) for the treatment of tinea pedis, heal cracks, calluses and dry feet.

SUMMARY:
A prospective, open post-market clinical investigation that will enroll male and female subjects diagnosed with foot fungus and at least one of the following conditions: heal cracks, calluses and/or dry feet. The investigation population will consist of 48 subjects fulfilling the eligibility criteria for the clinical investigation. The subjects will all be treated with the study product, Nåva Foot Cream. The duration of the investigation is estimated to 6 months, including a 2-month recruitment period and 2-month follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. > 18 years of age
3. Tinea pedis (Athlete's foot) confirmed with positive mycological culture for a dermatophyte
4. Total score of 6-16 when grading the eight sign and symptoms of tinea pedis (erythema, erosions, macerations, pruritus, fissures, burning/stinging, hyperkeratosis, odour) using a 4-point severity scale (0=absent, 1= mild, 2= moderate, 3=severe)

   o Score of 2 or higher required in at least one of the following: erythema, pruritus, macerations or odour
5. Score of at least 2 (moderate) required in at least one of the following: heel cracks (rhagades), calluses and dry feet (hyperkeratosis) using a 5-point severity scale (0=absent, 1= mild, 2= moderate, 3= advanced, 4=severe) age

Exclusion Criteria:

1. Patients with negative mycological culture
2. Severe tinea pedis interdigitalis (Athlete's foot) total score of grading sign and symptoms > 16
3. Women pregnant or lactation at time of enrolment
4. Patients using medicinal topical antifungal therapy within 4 weeks prior to study start
5. Treatment with oral terbinafine, itraconazole or fluconazole within 6 months prior to start of study
6. Treatment with other systemic antifungals within 12 weeks prior to start of study
7. Treatment with systemic corticosteroids or immunosuppressants within 6 weeks prior to start of study
8. Any other condition that as judged by the investigator may make follow-up or investigations inappropriate
9. Any patient that according to the Declaration of Helsinki is unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Effective clinical treatment rate | Baseline to end of study (8 weeks)
  Change of total mean score (TMS): Improvement of 8 clinical signs and symptoms of foot fungus calculated as the total score of all using a 4-point severity scale for each symptom.

SECONDARY OUTCOMES:
Frequency of negative fungal culture | Baseline to end of study (8 weeks)
  Frequency of patients with negative fungal culture at end of study.
Frequency of negative KOH test | Baseline to end of study (8 weeks)
  Frequency of patients with negative KOH test at end of study
Tolerability to the device used | Baseline to end of study (8 weeks)
  Tolerability assessed using a 5-point Likert scale (very good, good, moderate, poor, and very poor)
Other clinical signs and symptoms | Baseline to end of study (8 weeks)
  • Long term follow-up (8 weeks) on patient outcomes on heel cracks(rhagades), calluses and/or dry feet (hyperkeratosis)
Dermatology Quality of life | Baseline to end of study (8 weeks)
  Dermatology QoL Index

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lundvall, Principal Investigator — Region Örebro län
Locations (3):
- Sweden (3):
  - Carlanderska sjukhuset, Gothenburg
  - Univeristetssjukhuset, Örebro
  - PTC, Skövde

IPD SHARING:
Plan to Share IPD: No